CLINICAL TRIAL: NCT05778344
Title: Efficacy of Teletechnology-assisted Home-based Exercise Program for Severe COVID-19
Brief Title: Teletechnology-assisted Home-based Exercise Program for Severe COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, Mr. Ping-Lun Hsieh, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202106133RIND
Record Dates: First submitted 2023-03-13; First posted 2023-03-21 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: COVID-19; Telerehabilitation
Keywords: Pulmonary Rehabilitation
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-based pulmonary rehabilitation group (Experimental): The home-based pulmonary rehabilitation group received breathing exercise instructions using online learning materials soon after randomization. The participants received a home-based exercise plan, which comprised aerobic exercise and resistance exercise with instruction sheets. Teletechnology was incorporated into home-based pulmonary rehabilitation via videotelephony (or telephone calls if indicated). Time points for these teletechnology-assisted consultations were at day 7, day 14 after randomization and every 2 weeks after that until the completion of the study (week 12).
  Interventions: Behavioral: Teletechnology-assisted home-based pulmonary rehabilitation
- Usual care group (Active Comparator): The usual care group will receive breathing exercise instructions using online learning materials soon after randomization. The participants will also receive general exercise education and exercise safety principles but not any consultation about their physical activity/exercise during the study period.
  Interventions: Behavioral: Teletechnology-assisted home-based pulmonary rehabilitation

INTERVENTIONS:
Behavioral: Teletechnology-assisted home-based pulmonary rehabilitation — The accuracy and safety of home-based pulmonary rehabilitation will be checked regularly through technology devices such as smart watch and via videotelephony (or telephone calls if indicated).

SUMMARY:
The aim of this study was to investigate the efficacy of a home-based pulmonary rehabilitation program with the support of teletechnology in COVID-19 survivors. The main questions it aims to answer were:

* The change of six-minute walk distance
* The change of time of one-minute sit-to-stand test
* The change of maximal strength of upper-limb, lower-limb and respiratory muscle
* The change of quality of life Participants in the home-based pulmonary rehabilitation group received teletechnology-assisted consultations (either by videotelephony or telephone calls) for every 1-2 weeks during the intervention period, and participants in the usual care group did not receive teletechnology-assisted consultations during the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Patients are 20 years or more with severe (severe pneumonia) to critical (acute respiratory distress syndrome, sepsis, or septic shock) COVID-19 during hospitalization after deisolation.
* Patients are 65 years or more, or ever receiving oral antiviral treatment after deisolation.
* Patient have the ability to ambulate on level surface without direct contact of another person, have telecommunication device(s), and provide consent to receive teletechnology-assisted rehabilitation.

Exclusion Criteria:

* Patients are pregnant or planning for pregnancy.
* Patients have cognitive dysfunction, learning disability, uncontrolled arrhythmia or hypertension, or any medical diagnosis other than COVID-19 that would prominently influence their ability to follow instructions and perform exercise.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-04-12 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-05-24 (Actual)

PRIMARY OUTCOMES:
Six-minute walk distance | Week 0
  The distance of six-minute walk test
Six-minute walk distance | Week 4
  The distance of six-minute walk test
Six-minute walk distance | Week 8
  The distance of six-minute walk test
Six-minute walk distance | Week 12
  The distance of six-minute walk test
Six-minute walk distance | Week 24
  The distance of six-minute walk test

SECONDARY OUTCOMES:
Maximal upper limb strength | Week 0
  Hand grip strength
Maximal upper limb strength | Week 4
  Hand grip strength
Maximal upper limb strength | Week 8
  Hand grip strength
Maximal upper limb strength | Week 12
  Hand grip strength
Maximal upper limb strength | Week 24
  Hand grip strength
Maximal lower limb strength | Week 0
  Leg press strength
Maximal lower limb strength | Week 4
  Leg press strength
Maximal lower limb strength | Week 8
  Leg press strength
Maximal lower limb strength | Week 12
  Leg press strength
Maximal lower limb strength | Week 24
  Leg press strength
Maximal respiratory muscle strength | Week 0
  Inspiratory and expiratory pressure of respiratory muscle
Maximal respiratory muscle strength | Week 4
  Inspiratory and expiratory pressure of respiratory muscle
Maximal respiratory muscle strength | Week 8
  Inspiratory and expiratory pressure of respiratory muscle
Maximal respiratory muscle strength | Week 12
  Inspiratory and expiratory pressure of respiratory muscle
Maximal respiratory muscle strength | Week 24
  Inspiratory and expiratory pressure of respiratory muscle
Quality of life score | Week 0
  Quality of life assessed by Short-form 12 questionnaire
Quality of life score | Week 4
  Quality of life assessed by Short-form 12 questionnaire
Quality of life score | Week 8
  Quality of life assessed by Short-form 12 questionnaire
Quality of life score | Week 12
  Quality of life assessed by Short-form 12 questionnaire
Quality of life score | Week 24
  Quality of life assessed by Short-form 12 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ping-Lun Hsieh, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Felten-Barentsz KM, van Oorsouw R, Klooster E, Koenders N, Driehuis F, Hulzebos EHJ, van der Schaaf M, Hoogeboom TJ, van der Wees PJ. Recommendations for Hospital-Based Physical Therapists Managing Patients With COVID-19. Phys Ther. 2020 Aug 31;100(9):1444-1457. doi: 10.1093/ptj/pzaa114. PMID 32556323
- [Background] Gloeckl R, Leitl D, Jarosch I, Schneeberger T, Nell C, Stenzel N, Vogelmeier CF, Kenn K, Koczulla AR. Benefits of pulmonary rehabilitation in COVID-19: a prospective observational cohort study. ERJ Open Res. 2021 May 31;7(2):00108-2021. doi: 10.1183/23120541.00108-2021. eCollection 2021 Apr. PMID 34095290
- [Background] Betschart M, Rezek S, Unger I, Beyer S, Gisi D, Shannon H, Sieber C. Feasibility of an Outpatient Training Program after COVID-19. Int J Environ Res Public Health. 2021 Apr 9;18(8):3978. doi: 10.3390/ijerph18083978. PMID 33918887